CLINICAL TRIAL: NCT03096782
Title: Cord Blood Ex-Vivo MSC Expansion Plus Fucosylation to Enhance Homing and Engraftment
Brief Title: Umbilical Cord Blood Transplant With Added Sugar and Chemotherapy and Radiation Therapy in Treating Patients With Leukemia or Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0051; NCI-2018-01236 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0051 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-03-21; First posted 2017-03-30 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Biphenotypic Leukemia; Acute Leukemia; Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Chemotherapy-Related Leukemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Myelomonocytic Leukemia; Hodgkin Lymphoma; Langerhans Cell Histiocytosis; Minimal Residual Disease; Myelodysplastic Syndrome; Myelodysplastic Syndrome With Excess Blasts; Non-Hodgkin Lymphoma; Recurrent Hodgkin Lymphoma; Refractory Acute Lymphoblastic Leukemia; Refractory Myelodysplastic Syndrome; Small Lymphocytic Lymphoma; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Hodgkin Disease; Histiocytosis, Langerhans-Cell; Neoplasm, Residual; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Lymphoma, Non-Hodgkin | interventions — Antilymphocyte Serum; thymoglobulin; Busulfan; Clofarabine; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; Melphalan; Mycophenolic Acid; Rituximab; CT-P10; Tacrolimus; Whole-Body Irradiation; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemotherapy and Cord blood transfusion (Experimental): All patients received Busulfan as per standard of care. Busulfan test dose can be administered either as an outpatient prior to admission or as an inpatient on Day -10.
  Busulfan pharmacokinetics will be performed with the test dose and the first dose on Day -7 per standard of care. The doses of Days -6, -5, and -4 will be subsequently adjusted to target an AUC of 4,000 microMol.min-1. In the event that PK adjusting were not possible a dose of busulfan of 130 mg/m2 will be administered.
  GVHD PROPHYLAXIS: All patients also receive mycofenolate mofetil IV over 2 hours or PO BID on days -3 with a taper beginning on day 100 in the absence of GVHD, tacrolimus IV or PO starting on day -2 for 6 months in the absence of GVHD, and filgrastim-sndz SC QD starting on day 0 until white blood count begins to recover.
  Interventions: Biological: Anti-Thymocyte Globulin; Drug: Busulfan; Drug: Clofarabine; Drug: Cyclophosphamide; Biological: Filgrastim-sndz; Drug: Fludarabine; Drug: Melphalan; Drug: Mycophenolate Mofetil; Biological: Rituximab; Drug: Tacrolimus; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Clofarabine — Given IV
  Other Names: Clofarex; Clolar
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Filgrastim-sndz — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Zarxio
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Tacrolimus — Given IV
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo total body irradiation
  Other Names: Total Body Irradiation; Whole-Body Irradiation
Procedure: Umbilical Cord Blood Transplantation — Undergo cord blood transplant
  Other Names: Cord Blood Transplantation; UCB transplantation

SUMMARY:
This phase II trial studies how well an umbilical cord blood transplant with added sugar works with chemotherapy and radiation therapy in treating patients with leukemia or lymphoma. Giving chemotherapy and total-body irradiation before a donor umbilical cord blood transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The umbilical cord blood cells will be grown ("expanded") on a special layer of cells collected from the bone marrow of healthy volunteers in a laboratory. A type of sugar will also be added to the cells in the laboratory that may help the transplant to "take" faster.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and feasibility of transplantation of cord blood which is expanded in mesenchymal precursor cell (MPC) co-cultures then fucosylated with fucosyltransferase (FT)-VI and guanosine diphosphate (GDP) fucose prior to infusion in patients with hematologic malignancies following high-dose therapy.

II. To evaluate the time to engraftment using expanded fucosylated cord blood.

SECONDARY OBJECTIVES:

I. To evaluate the rate and severity of graft versus host disease. II. To evaluate the rates of infectious complications. III. To evaluate the rates of disease-free and overall survival.

Summary: All patients receive Busulfan as per standard of care. Busulfan test dose can be administered either as an outpatient prior to admission or as an inpatient on Day -10.

Busulfan pharmacokinetics will be performed with the test dose and the first dose on Day -7 per standard of care. The doses of Days -6, -5, and -4 will be subsequently adjusted to target an AUC of 4,000 microMol.min-1. In the event that PK adjusting were not possible a dose of busulfan of 130 mg/m2 will be administered.

GVHD PROPHYLAXIS: All patients receive mycofenolate mofetil IV over 2 hours or orally (PO) twice daily (BID) on days -3 with a taper beginning on day 100 in the absence of GVHD, tacrolimus IV or PO starting on day -2 for 6 months in the absence of GVHD, and filgrastim-sndz subcutaneously (SC) once daily (QD) starting on day 0 until white blood count begins to recover.

After completion of study treatment, patients are followed up at months 1, 3, 6, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following hematologic malignancies: a. Acute myelogenous leukemia (AML), induction failure, high-risk for relapse first remission (with intermediate-risk or high-risk cytogenetics, flt3 mutation positive and/or evidence of minimal residual disease by flow cytometry), secondary leukemia from prior chemotherapy and/or arising from myelodysplastic syndrome (MDS), Langerhan's cell histiocytosis, any disease beyond first remission. b. Myelodysplastic syndrome (MDS): MDS International Prognostic Scoring System (IPSS) INT-1 will be enrolled only if the subjects have failed previous leukemia treatments and are transfusion-dependent. MDS may be primary or therapy related, including patients that will be considered for transplant. Including the following categories: 1) Revised IPSS intermediate and high risk groups, 2) MDS with transfusion dependency, 3) Failure to respond or progression of disease on hypomethylating agents, 4) Refractory anemia with excess of blasts, 5) Transformation to acute leukemia, 6) Chronic myelomonocytic leukemia, 7) Atypical MDS/myeloproliferative syndromes, 8) Complex karyotype, abn(3g), -5/5g-, -7/7g-, abn(12p), abn(17p). c. Acute lymphoblastic leukemia (ALL) patients with the following will be considered: induction failure, primary refractory to treatment (do not achieve complete remission after first course of therapy) or are beyond first remission including second or greater remission or active disease. Patients in first remission are eligible if they are considered high risk, defined as any of the following detected at any time: with translocations 9;22 or 4;11, hypodiploidy, complex karyotype, secondary leukemia developing after cytotoxic drug exposure, and/or evidence of minimal residual disease, or acute biphenotypic leukemia which excludes > 7 chromosomal abnormalities, or double hit non-Hodgkin's lymphoma. Non-Hodgkin's lymphoma (NHL) in second or third complete remission or relapse (including relapse post autologous hematopoietic stem cell transplant), or relapsed double hit lymphoma. Small lymphocytic lymphoma (SLL), or chronic lymphocytic leukemia (CLL) with progressive disease with progression after standard of care therapy or have failed/been intolerant to ibrutinib. Chronic myelogenous leukemia (CML) second chronic phase or accelerated phase. Hodgkin's disease (HD): Induction failure after the first complete remission, or relapse (including relapse post autologous hematopoietic stem cell transplant), or those with active disease.
* The first 6 patients must be >= 18 and =< 65 years old. The subsequent patients may include pediatric patients >= 12 and =< 65 years old. Eligibility for pediatric patients will be determined in conjunction with an MD Anderson Cancer Center (MDACC) pediatrician.
* Performance score of at least 80% by Karnofsky or performance score (PS) < 3 (Eastern Cooperative Oncology Group [ECOG]) (age >= 12 years)
* Left ventricular ejection fraction of > 40%.
* Pulmonary function test (PFT) demonstrating a diffusion capacity of least 50% predicted.
* Creatinine =< 1.5 mg/dL for patients 12 years old and older and =< 1 for patients younger than 12 years old.
* Serum glutamate pyruvate transaminase (SGPT) =< to 2.0 x normal.
* Bilirubin =< to 2.0 x normal.
* Negative beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization and willing to use an effective contraceptive measure while on study.
* Patients must have two cord blood (CB) units available which are matched with the patient at 4, 5, or 6/6 HLA class I (serological) and II (molecular) antigens. Each cord must contain at least 1.5 x 10^7 total nucleated cells/Kg recipient body weight (pre-thaw).
* Have identified a backup cells source in case of engraftment failure. The source can be autologous, related or unrelated.
* Patient must not have a 10/10 HLA matched family member or unrelated donor.
* Patients will have a back-up graft from any of the following: an available fraction of autologous marrow; or peripheral blood progenitor cells (PBPCs) harvested and cryopreserved; or family member donor; or a third cord blood unit.
* Prior to initiating chemotherapy in this study, twenty-one or more days must have elapsed since the patient's last radiation or chemotherapy administration (Hydrea, Gleevec and other tyrosine kinase inhibitors [TKI] as well as intrathecal therapy are accepted exceptions).

Exclusion Criteria:

* Patients with known history of human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS).
* Patients with positive hepatitis serology that is definitive of active disease.
* Active central nervous system (CNS) disease in patient with history of CNS malignancy.
* Patients with chronic active hepatitis or cirrhosis. If positive hepatitis serology, the study chair may deem the patient eligible based on the results of liver biopsy.
* Patients with uncontrolled serious medical condition such as persistent septicemia despite adequate antibiotic therapy, decompensated congestive heart failure despite cardiac medications or pulmonary insufficiency requiring intubation (excluding primary disease for which CB transplantation is proposed), or psychiatric condition that would limit informed consent.
* Positive beta HCG in female of child-bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization or breast-feeding.
* Pediatric patients with acute lymphoblastic leukemia (ALL) that is t (9,22) positive in first remission are not eligible unless there is evidence of minimal residual disease after initial induction and/or consolidation treatment or the pediatric Philadelphia chromosome positive (Ph+) ALL is clinically refractory to available therapies with evidence of persistence in the bone marrow or peripheral blood.
* Patients with options for treatment that are known to be curative are not eligible.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Olson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruitment from October 2017 to May 2022 at MD Anderson Cancer Center
Groups:
- Chemotherapy Plus Cord Blood Transplant: GVHD PROPHYLAXIS: All patients receive mycofenolate mofetil IV over 2 hours or PO BID on days -3 with a taper beginning on day 100 in the absence of GVHD, tacrolimus IV or PO starting on day -2 for 6 months in the absence of GVHD, and filgrastim-sndz SC QD starting on day 0 until white blood count begins to recover.
  Anti-Thymocyte Globulin: Given IV
  Busulfan: Given IV
  Clofarabine: Given IV
  Filgrastim-sndz: Given SC
  Fludarabine: Given IV
  Mycophenolate Mofetil: Given IV or PO
  Rituximab: Given IV
  Tacrolimus: Given IV
  Total-Body Irradiation: Undergo total body irradiation
  Umbilical Cord Blood Transplantation: Undergo cord blood transplant
Period: Overall Study
Arm/Group | Chemotherapy Plus Cord Blood Transplant
Started | 6
Completed | 4
Not Completed | 2
Not completed — Death | 1
Not completed — Participant Relapsed | 1

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy and Cord Blood Transfusion: All patients received Busulfan as per standard of care. Busulfan test dose can be administered either as an outpatient prior to admission or as an inpatient on Day -10.
  Busulfan pharmacokinetics will be performed with the test dose and the first dose on Day -7 per standard of care. The doses of Days -6, -5, and -4 will be subsequently adjusted to target an AUC of 4,000 microMol.min-1. In the event that PK adjusting were not possible a dose of busulfan of 130 mg/m2 will be administered.
  GVHD PROPHYLAXIS: All patients also receive mycofenolate mofetil IV over 2 hours or PO BID on days -3 with a taper beginning on day 100 in the absence of GVHD, tacrolimus IV or PO starting on day -2 for 6 months in the absence of GVHD, and filgrastim-sndz SC QD starting on day 0 until white blood count begins to recover.
  Anti-Thymocyte Globulin: Given IV
  Busulfan: Given IV
  Clofarabine: Given IV
  Cyclophosphamide: Given IV
  Filgrastim-sndz: Given SC
  Fludarabine: Given IV
  Melphalan: Given IV
  Mycophenolate Mofetil: Given IV or PO
  Rituximab: Given IV
  Tacrolimus: Given IV
  Total-Body Irradiation: Undergo total body irradiation
  Umbilical Cord Blood Transplantation: Undergo cord blood transplant
Arm/Group | Chemotherapy and Cord Blood Transfusion
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Engraftment
Description: Number of days from transplant when participants achieved engraftment measure by ANC of 0.5 for three consecutive days.
Time Frame: Up to 12 months after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Plus Cord Blood Transplant
Number analyzed (Participants) | 6
Participants
  Twenty Two Days | 2
  Twenty Nine Days | 1
  Thirty Days | 1
  Nine Days | 1
  Thirty Two Days | 1

2. Secondary Outcome: Disease-free Survival
Description: Number of participants that were in remission post transplant.
Time Frame: Up to12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Plus Cord Blood Transplant
Number analyzed (Participants) | 6
Participants
  Complete Remission at 30 days | 6
  Complete Remission at 12 months | 4

3. Secondary Outcome: Overall Survival
Description: Number of participants alive 1 year post transplant.
Time Frame: Up to 12 months after transplant
Population: One participant died 5 months post transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Plus Cord Blood Transplant
Number analyzed (Participants) | 5
Participants | 4

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to 12 months post-transplant. Serious and Other Adverse Events were monitored up to Day 100 post-transplant.
Arm/Group | Chemotherapy and Cord Blood Transfusion
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy and Cord Blood Transfusion (N=6)
Diarrhea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy and Cord Blood Transfusion (N=6)
Abdominal pain (Gastrointestinal disorders) | 1
Abnormal coagulopathy (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arm pain (Vascular disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
BK cystitis (General disorders) | 1
BK virus (General disorders) | 1
Blurry vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest tightness (Cardiac disorders) | 1
Chills (General disorders) | 2
CMV infection (Infections and infestations) | 1
Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Crackles to right lung (Respiratory, thoracic and mediastinal disorders) | 1
Deconditioning (General disorders) | 1
Decreased Appetite (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dry Eyes (Eye disorders) | 1
DVT (thrombosis) (Vascular disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Dysuria (Renal and urinary disorders) | 1
E. Coli pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Fluid Imbalance (General disorders) | 1
Fluid Overload (General disorders) | 1
Flu-like Symptoms (General disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Generalized body aches (General disorders) | 1
Hand-foot syndrome (General disorders) | 1
Headache (Nervous system disorders) | 3
Hematochezia (General disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
HHV6 infection (Infections and infestations) | 4
Hyperbilirubinemia (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1
Indigestion (dyspepsia) (Gastrointestinal disorders) | 1
Ingrown toenail (General disorders) | 1
Insomnia (Psychiatric disorders) | 3
Int elevated ALT (Renal and urinary disorders) | 1
Blurred Vision (Eye disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Lower back pain (Musculoskeletal and connective tissue disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Migraine (General disorders) | 1
Mucositis (Gastrointestinal disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Neuropathy (Nervous system disorders) | 2
Neutropenic fever (General disorders) | 3
Norovirus (General disorders) | 1
Parainfluenza URI (General disorders) | 1
Peripheral edema (General disorders) | 1
Platelet Infusion Reaction (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Tachycardia (Cardiac disorders) | 2
Urinary Tract Infection (BK virus) (Infections and infestations) | 3
Vaginal irritation (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 3
Weakness (Musculoskeletal and connective tissue disorders) | 1
Transaminitis (General disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Parainfluenza URI (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03096782/Prot_SAP_000.pdf